CLINICAL TRIAL: NCT05166304
Title: Rebamipide as an Adjunct to Methotrexate in Patients With Active Rheumatoid Arthritis
Brief Title: Rebamipide in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: October 6 University (Other)
Collaborators: Minia University, faculty of medicine (Unknown); Sohag University (Other)
Responsible Party: Principal Investigator, engy wahsh, lecturer of clinical pharmacy, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUFMIRB App N. 1007/12/2023
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — rebamipide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): patients will receive the standard therapy (methotrexate) plus placebo tablets
  Interventions: Drug: Placebo
- rebamipide (Experimental): 100 mg rebamipide taken orally daily plus Methotrexate 15 mg weekly
  Interventions: Drug: Rebamipide

INTERVENTIONS:
Drug: Rebamipide — patients will receive the standard therapy plus 100 mg Rebamipide three times daily
  Arms: rebamipide
Drug: Placebo — patients will receive the standard therapy (methotrexate) plus placebo tablets
  Arms: placebo

SUMMARY:
Although the aetiology of RA remains to be fully elucidated, interleukin (IL)-17 are believed to play a critical role in the pathogenesis of RA. Rebamipide is an antiulcer drug that protects gastric epithelial cells,improves gastric defense mechanisms by increasing gastric mucus. Rebamipide inhibited interleukin (IL)-17, also it inhibits IL-1β-induced RASF proliferation.

ELIGIBILITY:
Inclusion Criteria:

* patients with active rheumatoid arthritis (disease activity score-28 joints: DAS-28 > 3.2) based on the 2010 American College of Rheumatology (ACR) criteria16 were recruited.

rheumatoid Patients who received the standard therapy (i.e. one or more conventional DMARDs) for at least three months.

Exclusion Criteria:

1. History of biological DMARDS.
2. History of gastrointestinal surgery, GI ulceration,GI bleeding
3. Intolerance or allergy to rebamibide or methotrexate
4. Smoking or alcohol abuse
5. Any changes in using medication (changing the dosage or type of medicines)
6. Receive hormone replacement therapy, warfarin, and other anticoagulants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
ACR20 | at baseline and at week 12
  based on tender and swollen joint counts, patient's assessment of pain
Disease activity scale in 28 joints (DAS-28) | at baseline and at week 12
  Scale assessing severity of rheumatoid arthritis based on number of tender, swollen joints, erythrocyte sedimentation rate (ESR) levels, and patient self-assessment of his condition (global health assessment). Whereas "28" describes the number of different joints including in the measurement: proximal interphalangeal joints (10 joints), metacarpophalangeal joints (10), wrists (2), elbows (2), shoulders (2), knees (2).

SECONDARY OUTCOMES:
HAQ-DI (Health Assessment Score- Disability index) | at baseline and at week 12
  HAQ-DI (Health Assessment Score- Disability index), in which patients are asked to rate their capacity to perform 20 activities of daily living (ADL). Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section
CRP | at baseline and at week 12
  Serum level of C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Esraa Abdallah, Principal Investigator — Minia University; Engy Wahsh, Study Chair — October 6 University; Asmaa Elsayed, Study Director — Sohag University
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided